CLINICAL TRIAL: NCT06313008
Title: A Clinical Study Comparing Effects of Empagliflozin Versus Vildagliptin on Inflammatory Biomarkers, and Atrial Function in Coronary Artery Disease Patients With Type 2 Diabetes: EMBA-VILDA-Response Trial.
Brief Title: Empagliflozin Versus Vildagliptin in CAD Patients With T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMBA-VILDA-Response trial.
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease; Type 2 Diabetes
Keywords: CAD.; T2DM.; LVEF%.; Sortilin.; Empaglilozin.; Vildagliptin.
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — empagliflozin; Vildagliptin

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized, double-dummy, blinded-endpoint, parallel-group trial that enrolled 120 CAD patients with T2DM. The patients were randomized 1: 1 for 6 months administration of empagliflozin or vildagliptin.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental): Eligible subjects were randomly and equally assigned to the empagliflozin add-on group (empagliflozin 10 mg/ day).
  Interventions: Drug: Empagliflozin 10 MG
- Vildagliptin (Experimental): 60 patients recieved vildagliptin as add-on group (vildagliptin 50 mg/day as the initial dose).
  Interventions: Drug: Vildagliptin 50 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — eligible subjects were randomly and equally assigned to the empagliflozin add-on group (empagliflozin 10 mg/ day).
  Other Names: Empa
  Arms: Empagliflozin
Drug: Vildagliptin 50 MG — eligible subjects were randomly and equally assigned to vildagliptin add-on group (vildagliptin 50 mg/day as the initial dose).
  Other Names: Vilda
  Arms: Vildagliptin

SUMMARY:
We compared the cardioprotective effects of empagliflozin, an SGLT2 inhibitor, with those of vildagliptin, a dipeptidyl peptidase-4 (DPP-4) inhibitor, focusing on various inflammatory biomarkers lipid profile, and cardiac function, in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This was a prospective, randomized, double-dummy, parallel-group trial that enrolled 120 patients with T2DM. The patients were randomized 1: 1 for 6 months administration of empagliflozin or vildagliptin. by using consecutive ascending randomization numbers in the treatment blocks allocated to each study site. The randomization was stratified by the presence or absence of statin and oral antidiabetic therapy. The randomization list was produced using an automated random number generator.

Clinical parameters, assessment of atrial myocardial function, LVEF%, LA diameter, glycemic and lipid profile, adiponectin, high-sensitivity C-reactive protein, and Sortilin levels will be determined at baseline and after the 6 months of treatment period.

Patient compliance was evaluated by the counting of pills by a physician at selected time-points. In addition, patients were provided with individual diary cards to record administration of the study medication on a daily basis. These cards were checked regularly by site staff.

The study will be approved by the local ethics committee and was conducted in accordance with the Declaration of Helsinki and its amendments. All included patients provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. T2DM patients with chronic stable angina.
2. patients with glycated hemoglobin (HbA1c) levels of 6.0-10.0%.
3. patients aged 20-80 years.
4. patients with a body mass index of ≥ 22 kg/m2.
5. patients who provided written informed consent.

Exclusion Criteria:

1. patients with type 1 diabetes mellitus or secondary diabetes mellitus.
2. patients with renal dysfunction (estimated glomerular filtration rate < 45 mL/min/1.73 m2).
3. patients with left ventricular ejection fraction (LVEF) < 30%.
4. patients with untreated cancer.
5. patients with hepatic cirrhosis.
6. patients with liver failure that was virus-, autoimmune- or drug-induced.
7. patients with alcoholism.
8. pregnant or breastfeeding patients, or those planning to become pregnant during the course of the study.
9. patients allergic to empagliflozin or vildagliptin.
10. patients with anemia (hemoglobin < 12 g/dL).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
LVEF % | 6 months
  echocardiographic measurements
Sortilin (ng/ml) | 6 months
  Serum Biomarkers
LDL (mg/dl) | 6 months
  Lipid profile

SECONDARY OUTCOMES:
hsCRP (mg/L) | 6 months
  Serum Biomarkers
HbA1c % | 6 months
  Glycemic control
FBG (mg/dl) | 6 Months
  Serum level

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Khedr, Prof., Study Director — Tanta University
Locations (1):
- Rehab Hussein Werida, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanaka A, Shimabukuro M, Okada Y, Taguchi I, Yamaoka-Tojo M, Tomiyama H, Teragawa H, Sugiyama S, Yoshida H, Sato Y, Kawaguchi A, Ikehara Y, Machii N, Maruhashi T, Shima KR, Takamura T, Matsuzawa Y, Kimura K, Sakuma M, Oyama JI, Inoue T, Higashi Y, Ueda S, Node K; EMBLEM Trial Investigators. Rationale and design of a multicenter placebo-controlled double-blind randomized trial to evaluate the effect of empagliflozin on endothelial function: the EMBLEM trial. Cardiovasc Diabetol. 2017 Apr 12;16(1):48. doi: 10.1186/s12933-017-0532-8. PMID 28403850
- [Background] Shimizu W, Kubota Y, Hoshika Y, Mozawa K, Tara S, Tokita Y, Yodogawa K, Iwasaki YK, Yamamoto T, Takano H, Tsukada Y, Asai K, Miyamoto M, Miyauchi Y, Kodani E, Ishikawa M, Maruyama M, Ogano M, Tanabe J; EMBODY trial investigators. Effects of empagliflozin versus placebo on cardiac sympathetic activity in acute myocardial infarction patients with type 2 diabetes mellitus: the EMBODY trial. Cardiovasc Diabetol. 2020 Sep 25;19(1):148. doi: 10.1186/s12933-020-01127-z. PMID 32977831
- [Background] Schernthaner G, Schernthaner-Reiter MH, Schernthaner GH. EMPA-REG and Other Cardiovascular Outcome Trials of Glucose-lowering Agents: Implications for Future Treatment Strategies in Type 2 Diabetes Mellitus. Clin Ther. 2016 Jun;38(6):1288-1298. doi: 10.1016/j.clinthera.2016.04.037. Epub 2016 May 19. PMID 27210264
- [Background] Naing S, Poliyedath A, Khandelwal S, Sigala T. Impact of EMPA-REG OUTCOME(R) on the management of type 2 diabetes mellitus: a review for primary care physicians. Postgrad Med. 2016 Nov;128(8):822-827. doi: 10.1080/00325481.2016.1245093. Epub 2016 Oct 25. PMID 27701934